CLINICAL TRIAL: NCT00234572
Title: Phase II, Multicentre, Randomized, Double-blind Study in Acromegalic Patients Evaluating the Efficacy and Safety of a Single Deep Subcutaneous Administration of Lanreotide Autogel (60, 90 or 120mg) Versus Placebo Followed by a Single Blind Fixed Dose Phase Evaluating the Pharmacokinetic, Pharmacodynamic, Efficacy and Safety Profile of Multiple Deep Subcutaneous Administrations of Lanreotide Autogel (60, 90 & 120mg) Ending in Open Label Dose Titration Phase.
Brief Title: Efficacy and Safety Study of Varying Doses of Lanreotide Autogel in Patients With Acromegaly
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-28-52030-717
Record Dates: First submitted 2005-10-06; First posted 2005-10-07 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — lanreotide

INTERVENTIONS:
Drug: Lanreotide (Autogel formulation)

SUMMARY:
The purpose of this study is to compare the effectiveness of lanreotide autogel to placebo after a single injection. Effectiveness and safety were then also assessed following four fixed-dose injections and after one year of treatment given at titrated doses.

ELIGIBILITY:
Inclusion Criteria:

* documentation of a diagnosis of active acromegaly based on either of the following definitions:

  1. the patient has never received somatostatin analog nor dopaminergic agonist or had previously received this medication but had stopped more than 3 months before visit 1 and had a mean growth hormone (GH)level >5ng/mL at visit 1; or
  2. the patient was receiving treatment with a somatostatin analog (other than lanreotide autogel) or a dopaminergic agonist at visit 1, had a mean GH >3ng/mL at visit 2 (or visit 2a) and had at least a 100% increase in mean GH levels between visit 1 and visit 2 (or visit 2a)

Exclusion Criteria:

* receipt of radiotherapy for acromegaly within 3 years
* pituitary surgery within 3 months prior to visit 1
* prior receipt of lanreotide autogel or GH antagonist
* anticipated need for pituitary surgery (adenomectomy) or radiotherapy during the study period
* known hypersensitivity to any of the test materials or related compounds
* clinically significant renal or hepatic abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2000-05; Primary Completion 2003-01-03 (Actual); Study Completion 2003-01-03 (Actual)

PRIMARY OUTCOMES:
Mean serum GH levels determined from serial measurements at screening, weeks 4, 13, 14, 15, 16, 32 & 52, and in the event of early withdrawal

SECONDARY OUTCOMES:
Serum IGF-1 levels determined at screening, at weeks 4, 13, 14, 15, 16, 32 & 52, and in the event of early withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (29):
- United States (11):
  - Baptist Health System Inc, Birmingham, Alabama
  - Pituitary Center, Los Angeles, California
  - Northwestern Medical Facility, Chicago, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - New York University Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Ben Taub Hospital, Houston, Texas
- Czechia (3):
  - St Ann's Faculty Hospital, Brno
  - University Hospital Charles University, Hradec Králové
  - Charles University, Prague
- France (4):
  - Clinique Marc Linquette, Lille
  - Hôpital Lariboisière - Service de Médecine B, Paris
  - Hôpital Cochin - Service d'Endocrinologie, Paris
  - CHRU de Brabois, Vandœuvre-lès-Nancy
- Germany (3):
  - Universitätklinikum Charité, Berlin
  - Med. Klinik der Universitätat Essen, Essen
  - Medizinische Klinik Innenstadt, München
- Queen Mary Hospital, Pokfulam, Hong Kong
- Hungary (2):
  - Semmelweiss University Medical School, Budapest
  - Semmelweiss University, Budapest
- Netherlands (2):
  - Academic Hospital Leiden, Leiden
  - Academic Hospital Rotterdam, Rotterdam
- United Kingdom (3):
  - Queen Elizabeth Hospital, Edgbaston, Birmingham
  - The Royal Free Hospital, Hampstead, London
  - Christie Hospital, Manchester

REFERENCES:
- [Result] Melmed S, Cook D, Schopohl J, Goth MI, Lam KS, Marek J. Rapid and sustained reduction of serum growth hormone and insulin-like growth factor-1 in patients with acromegaly receiving lanreotide Autogel therapy: a randomized, placebo-controlled, multicenter study with a 52 week open extension. Pituitary. 2010;13(1):18-28. doi: 10.1007/s11102-009-0191-1. Epub 2009 Jul 29. PMID 19639415